CLINICAL TRIAL: NCT04403022
Title: A Prospective, Multi-Center Investigation of the da Vinci SP® Surgical System in Colorectal Procedures for Benign and Malignant Disease
Brief Title: da Vinci SP® Investigational Device Exemption Study in Colorectal Procedures
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: dV SP - CR-01
Record Dates: First submitted 2020-05-14; First posted 2020-05-27 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Colorectal Cancer; Benign or Malignant Rectal or Colon Tumors
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — Robotic Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Single arm (Other): Colorectal procedure will be performed by da Vinci SP® Surgical System
  Interventions: Device: Robotic Assisted Surgery

INTERVENTIONS:
Device: Robotic Assisted Surgery — da Vinci SP Surgical System, instruments, and accessories in complex colorectal procedures such as low anterior resection procedure or right colectomy with or without total mesorectal excision

SUMMARY:
To confirm the safety and performance of the da Vinci SP Surgical System, Instruments and Accessories in a complex colorectal procedure such as low anterior resections or right colectomy.

DETAILED DESCRIPTION:
Primary Performance:

* The primary performance endpoint will be assessed as the ability to complete the planned da Vinci SP-assisted colorectal procedure without conversion to an alternate approach. Conversion* to an alternate approach comprises conversion to open, multiport laparoscopic**, multiport robotic or hand-assisted§ approach requiring undocking of the da Vinci SP Surgical System in order to complete the planned procedure using the alternate approach.

  * Performing an extracorporeal anastomosis is not considered a conversion ** Use of additional assistant laparoscopic port(s) is not considered a conversion § Laparoscopic or robotic with hand assistance

Primary Safety:

• The primary safety endpoint will be assessed as the incidence of all intraoperative and post-operative adverse events that occur through the 42-day follow-up period

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* BMI ≤ 35
* Candidate for single-port robotic-assisted surgery for low anterior resection with or without total mesorectal excision or right colectomy procedures
* ASA ≤ 3
* Willing and able to provide a written informed consent document
* Willing and able to comply with the study protocol requirements including perioperative follow-up examinations at 14 days, 42 days post operatively, and post-market long-term follow-up on an annual basis through 5 years

Exclusion Criteria:

* Clinical or radiological evidence of metastatic disease
* Life expectancy less than 6 months
* Cancer of the anal canal requiring an abdominoperineal resection
* Subjects with threatened mesorectal margins (≤1 mm) on MRI or ultrasound (for LAR ONLY)
* Subjects with planned major concomitant procedures (eg. hepatectomaies, other intestinal resections) or emergent case
* Subjects undergoing both LAR/TME and right colectomy during the same operation
* Preoperative colonoscopy demonstrating synchronous colorectal cancer
* History of inflammatory bowel disease
* Subject has a known bleeding or clotting disorder
* Uncontrolled illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Subject is contraindicated for general anesthesia or surgery
* Subject had prior incisional hernia with mesh repair
* Subject belongs to vulnerable population
* Subject is pregnant or suspected to be pregnant

Intraoperative Exclusion Criteria:

• Subject presents with adhesions or scarring in the pelvis which in the opinion of the investigator limits the ability to perform the minimally invasive procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-06-03 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Performance | IntraOperative period
  Performance defined as ability to complete the planned da Vinci SP-assisted colorectal procedure without conversion to an alternate approach.
Adverse Events Rates | Intraoperative through the 42-day postoperative period
  Safety defined as the incidence of all intraoperative and post-operative adverse events that occur through the 42-day follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Madhu L Gorrepati, Study Director — Clinical Affairs Director
Locations (9):
- United States (7):
  - Adventist Health System/Sunbelt, Orlando, Florida
  - Henry Ford, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - MountianView Hospital, Las Vegas, Nevada
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Houston Methodist Research Institute, Houston, Texas
  - MultiCare - Tacoma, Tacoma, Washington
- South Korea (2):
  - Ulsan University Hospital, Ulsan, Dong-gu
  - Ewha Womans University College of Medicine, Seoul, Gangseo-gu

IPD SHARING:
Plan to Share IPD: No